CLINICAL TRIAL: NCT00504530
Title: A Randomised, Double-blind, Placebo Controlled, Proof of Concept Study to Assess the Efficacy, Safety and Acceptability of r-hLIF for Improving Embryo Implantation Following in Vitro Fertilisation (IVF) and Embryo Transfer (ET) in Women With Recurrent Implantation Failure.
Brief Title: r-hLIF for Improving Embryo Implantation in IVF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Merck Serono International SA, an affiliate of Merck KGaA Darmstadt, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23079
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Infertility Implantation Failure
MeSH Terms: interventions — Leukemia Inhibitory Factor

INTERVENTIONS:
Drug: Emfilermin, recombinant human leukemia inhibitory factor (r-hLIF)

SUMMARY:
This study was designed to obtain pilot clinical evidence of the efficacy, safety and acceptability of r-hLIF administered during the luteal phase after IVF/intra-cytoplasmic sperm injection (ICSI) and ET for improving embryo implantation in infertile women with a history of at least three implantation failures following ART. Based on LIF expression patterns and experimental data from animal research a role of LIF in embryo implantation is anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal woman aged 21 to 36 years, inclusive, at time of consent
2. Infertile woman who justified IVF-ET or ICSI-ET treatment and who wished to conceive
3. A history of at least three ART cycles resulting in a transfer of at least two apparently healthy embryos and no evidence of implantation menstruation and/or beta hCG < 10 IU/L at the end of the cycle)
4. Had regular ovulatory spontaneous menstrual cycles lasting 25 to 35 days
5. Had FSH assessment (early follicular day 2 to 5) within the past six months < 12 IU/L
6. No other diagnosed cause of previous ART failure other than recurrent implantation failure
7. A body mass index (BMI) of ³ 20 and £ 30 kg/m2, calculated according to the following formula: BMI (kg/m2) = Body Weight (kg) / Height * Height (m2)
8. The presence of both ovaries
9. A uterine cavity without abnormalities which, in the investigator's opinion, could impair embryo implantation or pregnancy outcome, as assessed by ultrasound (US) examination performed within six months prior to beginning GnRH-agonist therapy
10. Normal cervical cytology within three years prior to beginning GnRH- agonist therapy.
11. At least one wash-out cycle (defined as ³ 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment, prior to beginning GnRH-agonist therapy
12. Male partner semen analysis within the six months prior to starting GnRH agonist therapy
13. Had a negative pregnancy test (urinary) within seven days of commencing GnRH-agonist therapy.
14. Willingness and ability to comply with the protocol for the duration of the study
15. Written informed consent given prior to any study related procedure not part of the patient's normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Known to be positive for Human Immunodeficiency Virus
2. Known to be positive for Hepatitis B or C Virus
3. Known allergy to E. coli derived pharmaceutical product
4. Any clinically significant systemic disease (e.g. insulin-dependant diabetes mellitus, epilepsy, severe migraine, intermittent porphyria, hepatic, renal or cardiovascular disease, severe corticosteroid-dependent asthma) or any significant allergic disease (excluding rhinitis, hay fever or sinusitis of ENT origin)
5. Presence of an uncontrolled clinically significant medical condition (including infection) as determined by the investigator
6. Persistent tachycardia defined as heart rate > 90 bpm confirmed by ECG
7. Any medical condition, which in the judgement of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug. In case of doubt, the patient in question was to be discussed with Serono's Study Director
8. More than one previous failed ART cycle, where "failed" is defined as cancellation of administration of hCG due to a poor response to gonadotrophin stimulation (defined as retrieval of three oocytes or less)
9. Any history of difficulties in ET procedure (i.e. requiring general anaesthetic e.g. due to position of cervix)
10. Hyperprolactinaemia, defined as prolactin levels of ³ 1000 mIU/L and/or the patient remained anovulatory despite appropriate dopamine agonist treatment
11. Abnormal undiagnosed gynaecological bleeding
12. Any contraindication to being pregnant and/or carrying pregnancy to term
13. Presence of any medical condition for which the use of gonadotrophin preparations or progesterone was contra-indicated
14. Known allergy or hypersensitivity to gonadotrophin preparations
15. Known intolerance or allergy to paracetamol (acetaminophen)
16. Active substance abuse
17. Previous entry into this study or simultaneous participation in another clinical drug trial

Ages: 21 Years to 36 Years | Sex: Female
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2001-09; Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Improvement of embryo implantation and Safety | Various

SECONDARY OUTCOMES:
Secondary endpoints were implantation rate, proportion of patients with biochemical pregnancy and the number of live births. | various

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brinsden, M.D., Principal Investigator — Bourn Hall Clinic, Bourn Hall, High Street, Bourn, Cambridge CB3 7TR

REFERENCES:
- [Result] Paterson JM, Smith SM, Simpson J, Grace OC, Sosunov AA, Bell JE, Antoni FA. Characterisation of human adenylyl cyclase IX reveals inhibition by Ca(2+)/Calcineurin and differential mRNA plyadenylation. J Neurochem. 2000 Oct;75(4):1358-67. doi: 10.1046/j.1471-4159.2000.0751358.x. PMID 10987815